CLINICAL TRIAL: NCT01012271
Title: Diagnostic Accuracy of Direct MR Arthrography Of The Wrist At 1.5, 3.0 And 7.0T
Status: Completed | Type: Observational
Sponsor: University of Zurich (Other)
Responsible Party: Principal Investigator, Gustav Andreisek, mg, University of Zurich
Other Study IDs: 002
Record Dates: First submitted 2009-11-11; First posted 2009-11-13 (Estimated); Last update posted 2016-03-30 (Estimated); Status verified 2016-03

CONDITIONS: Wrist Injuries
Keywords: Wrist abnormalities
MeSH Terms: conditions — Wrist Injuries

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

INTERVENTIONS:
Other: MRI — MR arthrography is used to evaluate wrist abnormalities

SUMMARY:
The purpose of our study is to evaluate the diagnostic accuracy of MR arthrography of the wrist at 1.5, 3.0, and 7.0T with wrist arthroscopy as reference standard.

ELIGIBILITY:
Inclusion criteria:

* age >18;
* clinical evidence for wrist joint abnormalities;
* request for MR arthrography prior to wrist arthroscopy;
* willingness to take part in our study with written informed consent;

Exclusion criteria:

* age<18;
* history of prior wrist surgery; systemic diseases e.g. rheumatoid arthritis;
* infection; history of adverse contrast reactions;
* contraindication for MR imaging (e.g. pacemaker, metallic implants, etc.);
* history or possible signs of renal failure (see section "nephrogenic systemic fibrosis")

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: primary care clinic
Sampling Method: Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2010-10; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: 01 Studienregister MasterAdmins, Study Director — UniversitaetsSpital Zuerich
Locations (1):
- Zurich, Switzerland